CLINICAL TRIAL: NCT06751017
Title: A Phase 1 Study to Assess the Effect of Carbamazepine on the Pharmacokinetics of S-892216 in Healthy Adult Participants
Brief Title: A Drug-drug Interaction Study of S-892216 Coadministered With Carbamazepime to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2315T1612
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: S-892216; Carbamazepine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Carbamazepine

STUDY DESIGN:
Intervention Model Description: 1-sequence, drug-drug interaction study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S-892216 (Experimental): Participants will receive S-892216 and carbamazepine.
  Interventions: Drug: S-892216; Drug: Carbamazepine

INTERVENTIONS:
Drug: S-892216 — S-892216 will be administered orally as a tablet.
Drug: Carbamazepine — Carbamazepine will be administered orally as a tablet.
  Other Names: Tegretol

SUMMARY:
The primary objective of this study is to investigate the effect of multiple-dose administration of carbamazepine on the pharmacokinetics of S-892216 in healthy adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Overtly healthy as determined by medical evaluation including medical history, medical examination, laboratory tests, vital sign measurements, and 12-lead electrocardiogram, at screening and on admission or participants whose laboratory values exceed the institutional reference range but deemed not clinically significant by the investigator in consideration of safety.
* Body mass index ≥18.5 and ≤32.0 kilograms/meter squared.

Exclusion Criteria:

* This study will not enroll participants with Asian ancestry, defined as individuals who have 1 or more Asian grandparent, due to significant increase of risk for carbamazepine-related serious dermatologic reactions almost exclusively in these populations.
* Presence or history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, or ophthalmological (that is, increased intra-ocular pressure) disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data per the investigator's assessment.
* History of adverse hematologic reaction to any drug, or a history of bone marrow depression.
* History or family history of severe cutaneous reactions including toxic epidermal necrolysis and Stevens-Johnson Syndrome.
* Prior carbamazepine use that was discontinued for tolerability or adverse events, including a clinically significant decrease in platelets, white blood cells, or hemoglobin.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of S-892216 | Days 1 and 35 (2 hours predose, 30 minutes to 144 hours postdose)
Time to Maximum Plasma Concentration (Tmax) of S-892216 | Days 1 and 35 (2 hours predose, 30 minutes to 144 hours postdose)
Plasma Concentration of Carbamazepine | Day 35 (2 hours predose, 30 minutes to 24 hours postdose)
Tmax of Carbamazepine | Day 35 (2 hours predose, 30 minutes to 24 hours postdose)

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 49

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Lenexa, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No